CLINICAL TRIAL: NCT00214513
Title: Maintain. A Randomized Trial of Effect of Low-Cost Maintenance Training on Exercise Capacity, Quality of Life and Morbidity
Brief Title: A Randomized Trial of Effect of Low-Cost Maintenance Training on Exercise Capacity, Quality of Life and Morbidity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amager Hospital (Other)
Collaborators: Bispebjerg Hospital (Other); University of Copenhagen (Other); Danish Heart Foundation (Other); Ministry of the Interior and Health, Denmark (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Maintain
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2007-05-17 (Estimated); Status verified 2007-05

CONDITIONS: Chronic Heart Failure

INTERVENTIONS:
Behavioral: Home-based exercise training

SUMMARY:
The aim of the study is to determine whether a low-cost home-based training programme can maintain the achieved effect of physical training on exercise capacity and QOL in patients with Chronic Heart Failure.

DETAILED DESCRIPTION:
Guidelines recommend physical training in the treatment of patients with CHF. Several studies have demonstrated that even short-term training programmes can increase maximal oxygen intake, improve muscular strength, reduce neurohumoral activity and result in other effects, which are of potential benefit. Following 2-3 months training at 70 - 80% of maximal capacity, improved exercise capacity and oxygen uptake due to increased cardiac output and also better oxygen uptake in the peripheral muscles have been demonstrated. Moreover, studies have indicated an improvement of the quality of life (QOL). However, the effects of exercise training are rapidly lost without maintenance. Thus the crucial question is to identify a method to sustain the physical activity outside an expensive, enthusiastic and highly motivating protocol.

The aim of the study is to determine whether a low-cost home-based training programme can maintain the achieved effect of physical training on exercise capacity and QOL in patients with Chronic Heart Failure.

Comparison:

Patients fulfilling specified criteria for Chronic Heart Failure are randomised to either eight weeks with supervised group-based training (1.5 hrs.) twice a week followed by home-based training according to a specified protocol with supervised group-based training every 2 weeks (1,5 hrs), or to eight weeks with supervised training followed by usual care. During the whole period patients in both groups can contact the Heart Failure Clinic when needed.

ELIGIBILITY:
Inclusion Criteria:

1. NYHA II-IV
2. Ejection Fraction ≤45% assessed by echocardiography within the last 6 months
3. Optimal medical treatment according to guidelines
4. Informed consent -

Exclusion Criteria:

1. Hæmodynamically significant obstructive heart valve disease
2. Hæmodynamically significant valve insufficiency
3. Recent Myocardial infarction (8 weeks)
4. Significant arrythmia at exercise testing (NSVT, VT, VF or SVT with ventricular action >150)
5. Significant ischaemia or angina at low strain(£ 50 W)
6. Disabilities that render physical training impossible
7. Dementia
8. Serious other illness with expected shortened survival
9. Participation in other scientific protocols that do not allow participation
10. Lack of informed consent
11. If the patient cannot train in a team supervised by only one physiotherapist, e.g. due to poor balance, the patient can be excluded within the first two weeks of inclusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2004-06; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Primary endpoint: Exercise capacity based on standardised cycle ergometer test after 14 months.

SECONDARY OUTCOMES:
Secondary endpoints:
Maximum oxygen uptake at 14 months
Maximum exercise capacity measured by the Shuttle Walk test at 14 months
Exercise capacity measured by 6-minute walking test (6MWT)at 14 months
Muscular strength (sit-to-stand) at 14 months
QOL (SF36 and Minnesota) at 14 months
Serological tests including brain natriuretic peptide at 14 months
In a subgroup including 2x20 patients training-induced changes in muscle biopsies will be evaluated at 14 months.
After 1,3 and 5 years hospital-admissions and death through record linkage.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Prescott, MD, Principal Investigator — Dept of Cardiology, Rigshospitalet, Copenhagen, Denmark
Locations (1):
- Amager Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Prescott E, Hjardem-Hansen R, Dela F, Orkild B, Teisner AS, Nielsen H. Effects of a 14-month low-cost maintenance training program in patients with chronic systolic heart failure: a randomized study. Eur J Cardiovasc Prev Rehabil. 2009 Aug;16(4):430-7. doi: 10.1097/HJR.0b013e32831e94f8. PMID 19491687